CLINICAL TRIAL: NCT01636674
Title: Value of 18F-Fluordeoxyglucose Positron Emission Tomography/ Computed Tomography and Molecular Tumor Characterisation in Preoperative Staging og Postoperative Control of Colon Cancer
Brief Title: 18F-FDG PET/CT and Molecular Tumor Characterisation for Staging and Follow-up of Colon Cancer
Acronym: COLOPET1
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Naestved Hospital (Other)
Collaborators: University of Copenhagen (Other); Rigshospitalet, Denmark (Other); Region Zealand (Other)
Responsible Party: Principal Investigator, Bodil Elisabeth Engelmann, MD, research fellow, Naestved Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: SJ-82
Record Dates: First submitted 2012-07-06; First posted 2012-07-10 (Estimated); Last update posted 2012-07-10 (Estimated); Status verified 2012-07

CONDITIONS: Colon Cancer
Keywords: positron emission tomography; computed tomography; fluordeoxyglucose; colon cancer; cancer; staging; imaging
MeSH Terms: conditions — Colonic Neoplasms; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: 18F-fluordeoxyglucose positron emission tomography/ computed tomography — 18F-fluordeoxyglucose positron emission tomography/ computed tomography for preoperative staging and post-operative follow-up

SUMMARY:
The investigators are investigating the usefulness of 18F-Fluordeoxyglucose Positron Emission Tomography/ Computed Tomography (18F-FDG PET/CT) for staging and follow-up of colon cancer. Furthermore, the investigators combine 18F-FDG PET findings with clinical and histopathological features, circulating tumor cell (CTC) analyses, tumor gene expression and measurements of circulating cancer biomarkers sUPAR, TIMP-1 and CEA in order to predict tumor recurrence.

The investigators hypothesis: The combination of functional imaging by 18F-FDG PET/CT and pre-existing and evolving molecular biomarkers will optimize tumor characterization, staging of disease and early detection of recurrence.

ELIGIBILITY:
Inclusion Criteria:

* clinical or histological diagnosis of malignant clonic neoplasm (distance of more than 15 cm from anal ring)
* 18 years of age or older
* written informed consent

Exclusion Criteria:

* diabetes
* known malignant disease other than colon cancer
* known metastatic disease
* impairment of renal function
* allergy to CT contrast agents
* body weight of more than 150 kg
* claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2009-07; Primary Completion 2013-03 (Estimated); Study Completion 2013-03 (Estimated)

PRIMARY OUTCOMES:
time to recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Bodil E Engelmann, MD, Principal Investigator — Naestved Hospital